CLINICAL TRIAL: NCT01863901
Title: A Prospective, Non-Randomized, Unblinded Study Evaluating the Treatment With the Cryo-Touch III Device for Upper Limb Spasticity
Brief Title: Study Evaluating Treatment of Upper Limb Spasticity Using the Cryo-Touch III Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-0709
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Upper Limb Spasticity
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with the Cryo-Touch III Device (Experimental)
  Interventions: Device: Treatment with Cryo-Touch III device

INTERVENTIONS:
Device: Treatment with Cryo-Touch III device

SUMMARY:
A proof of concept study to evaluate the feasibility of safe and effective treatment of upper limb spasticity using the Cryo-Touch III Device.

DETAILED DESCRIPTION:
Spasticity, common in neurological disorders, is part of the upper motor neuron syndrome displaying increased tone, clonus, spasms, spastic dystonia and co- contractions. The impact of spasticity on the patient varies from a subtle neurological sign to severe spasticity causing pain and contractures. Upper limb spasticity (ULS) is the rapid contraction or shortening of the muscles in the arm causing abnormal muscle movements in the elbow, wrist and fingers. It has been reported that over 1 million Americans with traumatic injury to the brain or spinal cord, stroke, multiple sclerosis and cerebral palsy experience ULS. Tightly clenched fists, twisted wrist and elbow joints, and fixed arms in flexed positions result in extreme discomfort, pain and spasm. A nonsurgical, minimally invasive, effective approach to pain associated with ULS is desirable.

Myoscience, Inc. (Redwood City, CA) has developed a pain management device - the Cryo-Touch III - for a novel, minimally invasive procedure using focused cold therapy to target sensory nerve tissue and offer long-lasting pain relief through cryoanalgesia. The device operates on the well-established cryobiology principle that localized exposure to controlled, moderately low temperature conditions can alter tissue function. The therapy treats nerves via a probe in the form of an assembly of small diameter needles, creating a highly localized, low temperature treatment zone around the probe. This focused cold therapy creates a conduction block that prevents nerve signaling. Prior studies of the Cryo-Touch, Cryo-Touch II, Cryo-Touch III (a.k.a. PCP 1.0) devices have provided preliminary evidence of effectiveness on motor nerves and have been shown to be safe with no serious device-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and older.
2. Trial participants must have a confirmed diagnosis that results in spasticity involving muscle innervated by the musculocutaneous nerve (MCN).
3. Any medications must be maintained on a stable schedule for at least two weeks prior to treatment. No washout period is allowed.
4. Must have an average score on the Modified Ashworth Scale for Spasticity of ≥ 2 over the last 30 days in the elbow.
5. Subject, in the Investigator's opinion, will not be exposed to unacceptable risk by participation.

Exclusion Criteria:

1. Previous surgical intervention that altered the target neural anatomy of the upper limb.
2. Any injection (neurolytic, sclerosing, anesthetic, etc.) to the upper limb within the last 4 months.
3. Current enrollment in an investigational drug or device study that specifically targets spasticity management.
4. Allergy or intolerance to local anesthesia.
5. Any local skin condition at the treatment site that in the investigator's opinion would adversely affect treatment or outcomes.
6. Any chronic medication use (prescription, over-the-counter, etc.) that in the investigator's opinion would affect study participation or subject safety.
7. Diagnosis of cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, Raynaud's disease, open and/or infected wounds.
8. Diagnosis of progressive neurologic diseases such as ALS.
9. For any reason, in the opinion of the investigator, the subject may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, any related upper limb injury, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kansas City Bone and Joint Clinic, Overland Park, Kansas
  - Dr. Mitchell Paulin, Paoli, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for the study was initiated April 22, 2013 and was completed June 28, 2013 at two investigational sites.
Groups:
- Treatment With the Cryo-Touch III Device: Treatment with Cryo-Touch III device
Period: Overall Study
Arm/Group | Treatment With the Cryo-Touch III Device
Started | 19
Completed (Completion of Day 30 timepoint is considered a completed subject.) | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 19
Primary Diagnosis [Count of Participants; unit: Participants]
  Stroke | 16
  Traumatic Brain Injury | 2
  Other: Spinal Cord Injury | 1

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Pain and Symptoms Caused by Hypertonia in the Upper Arm as Measured by an Improvement of 1 Point or Greater on the Modified Ashworth Scale (MAS) at Day 7
Description: The Modified Ashworth Scale (MAS) is 6-point scale designed to assess muscle tone and spasticity through the flexion or extension of a joint. Muscle response is graded on a scale from 0 (no increase in muscle tone) to 4 (affected parts rigid in flexion or extension). This includes a 1+ rating, which further distinguishes the types of increase in muscle tone from those described by a 1 or 2 rating.
Time Frame: Baseline to: post-treatment (Day 0), Day 7, Day 30
Measure: Mean (Standard Deviation); unit: average MAS Score, absolute
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
average MAS Score, absolute
  Average MAS score Baseline | 3.3 (0.7)
  Average MAS score post-treatment | 1.3 (0.8)
  Average MAS Score Day 7 | 1.7 (0.9)
  Average MAS score Day 30 | 1.5 (0.9)

2. Secondary Outcome: Improvement in Spasticity as Measured by the Tardieu Scale
Description: The Tardieu Scale uses the application of stretch at several velocities to quantify muscle response and assess muscle spasticity. Two specified velocities were assessed (V1 and V2). For each stretch, quality of muscle reaction (X) is recorded on a 6-point scale from 0 (no resistance throughout passive movement) to 5 (immovable joint).
Time Frame: Baseline to: post-treatment (Day 0), Day 7, Day 30
Measure: Mean (Standard Deviation); unit: average X Score, absolute
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
average X Score, absolute
  Average X Score V1 Baseline | 1.7 (0.4)
  Average X score V1 at post-treatment | 1.1 (0.7)
  Average X Score V1 at Day 7 | 1.2 (0.7)
  Average X Score V1 at Day 30 | 0.8 (0.7)
  Average X Score V2 at Baseline | 1.9 (0.3)
  Average X score V2 post-treatment | 1.4 (0.7)
  Average X Score V2 at Day 7 | 1.5 (0.5)
  Average X Score V2 at Day 30 | 1.3 (0.7)

3. Secondary Outcome: Improvement in Spasm Frequency and Severity as Measured by the Penn Spasm Score
Description: The Penn Spasm Score, which is a patient reported score, consists of two sub-scales: the spasm frequency score and the spasm severity scale3. The Penn spasm frequency is assessed on a 5-point scale from 0 (no spasms) to 4 (spasms occurring more than ten times per hour). The spasm severity scale consists of three ratings, which are 1 (mild), 2 (moderate) and 3 (severe).
Time Frame: Baseline to: post-treatment (Day 0), Day 7, Day 30
Measure: Mean (Standard Deviation); unit: Average Penn Spasm Score, absolute
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
Average Penn Spasm Score, absolute
  Average Penn Frequency Score baseline | 1.3 (1.5)
  Average Penn Frequency Score Post-treatment | 0.7 (1.1)
  Average Penn Frequency Score Day 7 | 0.7 (1.1)
  Average Penn Frequency Score Day 30 | 0.7 (1.0)
  Average Penn Severity Score Baseline | 2.4 (0.5)
  Average Penn Severity Score Post-treatment | 1.6 (0.7)
  Average Penn Severity Score Day 7 | 1.8 (0.8)
  Average Penn Severity Score Day 30 | 2.1 (0.7)

4. Secondary Outcome: Improvement in Upper Extremity Motor Recovery as Measured by the Fugl-Meyer Scale (Post Stroke Subjects Only)
Description: The Fugl-Meyer Scale is an assessment consisting of 33 movements, each rated as "0" (cannot perform), "1" (can partially perform) or "2" (can perform fully). A Subject's score is the sum of their ratings on each of these items, where the maximum (best) score is a 66.
Time Frame: Baseline to: post-treatment (Day 0), Day 7, Day 30
Measure: Mean (Standard Deviation); unit: average Fugl-Meyer Sum Score, absolute
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 16
average Fugl-Meyer Sum Score, absolute
  Average Fugl-Meyer Sum Score Baseline | 24.5 (17.9)
  Average Fugl-Meyer Sum Score post-treatment | 27.3 (17.1)
  Average Fugl-Meyer Sum Score Day 7 | 24.6 (18.7)
  Average Fugl-Meyer Sum Score Day 30 | 22.3 (19.9)

5. Secondary Outcome: Subject Assessed Change in Mean Spasticity Numerical Rating Scale (NRS) Score
Description: The NRS is an 11-point scale from 0 to 10, where lower scores represent less spasticity.
Time Frame: baseline to: post-treatment (Day 0), Day 7, Day 30
Measure: Mean (Standard Deviation); unit: average NRS score, absolute
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
average NRS score, absolute
  average NRS Score baseline | 6.7 (2.0)
  Average NRS score post-treatment | 2.7 (1.5)
  Average NRS score Day 7 | 3.5 (1.6)
  Average NRS score Day 30 | 4.2 (1.8)

6. Secondary Outcome: Improvement in Pain as Assessed by Visual Analog Scale (VAS)
Description: Visual Analog Scale assesses pain on a 0-10 point range. 0= no pain and 10 is the worst pain imaginable. Higher score is associated with a worse outcome.
Time Frame: Baseline to: Post-treatment (Day 0), Day 7, Day 30
Measure: Mean (Standard Deviation); unit: average VAS Score, absolute
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
average VAS Score, absolute
  Average VAS score baseline | 1.0 (2.0)
  Average VAS score Post-treatment | 0.4 (0.8)
  Average VAS score Day 7 | 0.6 (1.4)
  Average VAS score Day 30 | 1.2 (2.1)

7. Secondary Outcome: Duration of Treatment Effect
Description: Subjects were asked to report the duration of treatment effect at Day 7,Day 30, and Day 56. Subjects could designate their results as "effect" "no effect" or "no longer effective". Subjects reporting "effect" at Day 56 were followed to Day 84; those with effect at Day 84 continued to be followed to Day 112.
Time Frame: Day 7, Day 30, Day 56, Day 84, Day 112
Population: Subjects reporting "effect" at Day 56 were followed to Day 84; those with effect at Day 84 continued to be followed to Day 112.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With the Cryo-Touch III Device
Number analyzed (Participants) | 19
Participants
  Day 7 | 15
  Day 30 | 17
  Day 56: number analyzed (Participants) | 17
  Day 56 | 10
  Day 84: number analyzed (Participants) | 10
  Day 84 | 7
  Day 112: number analyzed (Participants) | 7
  Day 112 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 0-Treatment day to Day 56-EOS.
Arm/Group | Treatment With the Cryo-Touch III Device
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With the Cryo-Touch III Device (N=19)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cellulitis right side of scrotum and groin (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With the Cryo-Touch III Device (N=19)
Soreness at triceps, left elbow (Musculoskeletal and connective tissue disorders) | 1 (1)
temporary increase in spasticity of treated extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
edema left clavicular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2012-11-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT01863901/Prot_000.pdf